CLINICAL TRIAL: NCT06251726
Title: Personalized Medicine in Early Stage Colorectal Cancer: Organ Preservation and Immune Benefit
Acronym: COLOSAVE
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Cancer Institute, France (Other Government); Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: APHP210349; PRT-K20-080 (Other Grant/Funding Number: French ministry of Health); 2021-018 (Other Grant/Funding Number: French National Cancer Institute)
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer
Keywords: Immunoscore; Tumor biomarkers; Organ preservation; Endoscopic submucosal dissection
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort of patients with stage T1 CRC treated by primary endoscopic resection.: Secondary surgery is performed in patients with pejorative histopathologic feature(s) of the tumor.
  Interventions: Diagnostic Test: Immunoscore Colon Test

INTERVENTIONS:
Diagnostic Test: Immunoscore Colon Test — Immunoscore Colon is an in-vitro diagnostic test, allowing the quantification of CD3 and CD8 positive cells in formalin-fixed paraffin-embedded (FFPE) tissue samples of primary colon cancer.
  The test uses immunohistochemistry, digital pathology techniques and a dedicated image analysis software to determine CD3+ and CD8 + cell densities in the tumor ant in the invasive margin of the tumor.

SUMMARY:
The overall aim of this study is to determine whether the Immunoscore associated with histopathological features of endoscopically resected stage T1 colorectal tumors is predictive of locoregional lymph node invasion, in order to better select patients eligible for an organ preservation strategy.

DETAILED DESCRIPTION:
The frequency of stage T1 superficial colorectal cancer (CRC) is around 15% and its incidence increases. In France, T1 superficial CCR is mostly treated with endoscopic submucosal dissection (ESD), offering potentially curative, organ-preserving treatment. The presence of pejorative histological criteria (eg. poor differentiation, budding, lymphovascular invasion), detected in about 50% of the tumors, leads to a secondary colectomy or rectal resection with postoperative complications and significant digestive, urological, and sexual functional sequelae. Strikingly, secondary surgical resection is performed in excess in 70 to 80% of the cases, given that no tumor is evidence in the colon and draining lymph nodes. Organ preservation (no secondary surgery) could be offered to a larger number of patients if biomarkers could complete the histological evaluation to better predict metastatic extension to lymph nodes.

Our team showed that the type, density, and location of immune cells in CRC strongly correlated with patients' survival at all disease stages. Our team created an "Immunoscore" (IS) assay, based on CD3+ and cytotoxic CD8+ T-cell densities determined by digital pathology in the tumor and its invasive margin. The robustness and prognostic performance of IS was validated in CRC . Sub-analysis of T1 tumors was not possible (only 31 cases) and tumor specimens did not result from endoscopic resection.

The objective of the study is to determine whether the Immunoscore associated with histopathological features of endoscopically resected stage T1 colorectal tumors is predictive of locoregional lymph node invasion, in order to better select patients eligible for an organ preservation strategy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old)
* patient with Stage T1 colorectal tumor
* treated by endoscopic resection between 2014 and 2019 in one of the participating sites
* sample of the resected tumor available for central analysis

Exclusion Criteria:

* Other Synchronous cancer
* Synchronous CRC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: French multi-institutional cohort of patients with stage T1 CRC treated by primary endoscopic resection
Sampling Method: Non-Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Lymph node invasion rate | time of histological examination of the surgical specimen
  Impact of Immunoscore stratification on lymph node invasion rate in patients with secondary surgery

SECONDARY OUTCOMES:
Lymph node invasion rate | time of histological examination of the surgical specimen
  Impact of Immunoscore stratification combined to Histological risk factors on lymph node invasion rate
Microenvironnement Immunologic parameters | Up to 3 years
  Assessment of Immunological features measured by RNA sequencing on tumor samples.
Molecular profile of the tumor | Up to 3 years
  Assessment of molecular profile of the tumor by transcriptomic profile measured by RNAseq. CMS classification will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Franck Pagès, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP - hôpital européen Georges-Pompidou, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol could be shared for the purpose of a metaanalysis.
Supporting Information: Study Protocol
Time Frame: One year after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI concerned. Teams wishing to obtain IPD must meet the sponsor and PI team to present their purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization.
  If all or part of the database is shared with countries outside the European Union for a future purpose, the contract between the sponsor and the recipient of the data that will guaranty levels of protection at least equivalent to those provided by EU regulation.

REFERENCES:
- [Background] Pages F, Mlecnik B, Marliot F, Bindea G, Ou FS, Bifulco C, Lugli A, Zlobec I, Rau TT, Berger MD, Nagtegaal ID, Vink-Borger E, Hartmann A, Geppert C, Kolwelter J, Merkel S, Grutzmann R, Van den Eynde M, Jouret-Mourin A, Kartheuser A, Leonard D, Remue C, Wang JY, Bavi P, Roehrl MHA, Ohashi PS, Nguyen LT, Han S, MacGregor HL, Hafezi-Bakhtiari S, Wouters BG, Masucci GV, Andersson EK, Zavadova E, Vocka M, Spacek J, Petruzelka L, Konopasek B, Dundr P, Skalova H, Nemejcova K, Botti G, Tatangelo F, Delrio P, Ciliberto G, Maio M, Laghi L, Grizzi F, Fredriksen T, Buttard B, Angelova M, Vasaturo A, Maby P, Church SE, Angell HK, Lafontaine L, Bruni D, El Sissy C, Haicheur N, Kirilovsky A, Berger A, Lagorce C, Meyers JP, Paustian C, Feng Z, Ballesteros-Merino C, Dijkstra J, van de Water C, van Lent-van Vliet S, Knijn N, Musina AM, Scripcariu DV, Popivanova B, Xu M, Fujita T, Hazama S, Suzuki N, Nagano H, Okuno K, Torigoe T, Sato N, Furuhata T, Takemasa I, Itoh K, Patel PS, Vora HH, Shah B, Patel JB, Rajvik KN, Pandya SJ, Shukla SN, Wang Y, Zhang G, Kawakami Y, Marincola FM, Ascierto PA, Sargent DJ, Fox BA, Galon J. International validation of the consensus Immunoscore for the classification of colon cancer: a prognostic and accuracy study. Lancet. 2018 May 26;391(10135):2128-2139. doi: 10.1016/S0140-6736(18)30789-X. Epub 2018 May 10. PMID 29754777
- [Background] Mlecnik B, Lugli A, Bindea G, Marliot F, Bifulco C, Lee JJ, Zlobec I, Rau TT, Berger MD, Nagtegaal ID, Vink-Borger E, Hartmann A, Geppert CI, Kolwelter J, Merkel S, Grutzmann R, Van den Eynde M, Jouret-Mourin A, Kartheuser A, Leonard D, Remue C, Wang J, Bavi P, Roehrl MHA, Ohashi PS, Nguyen LT, Han S, MacGregor HL, Hafezi-Bakhtiari S, Wouters BG, Masucci GV, Andersson EK, Zavadova E, Vocka M, Spacek J, Petruzelka L, Konopasek B, Dundr P, Skalova H, Nemejcova K, Botti G, Tatangelo F, Delrio P, Ciliberto G, Maio M, Laghi L, Grizzi F, Fredriksen T, Buttard B, Lafontaine L, Maby P, Majdi A, Hijazi A, El Sissy C, Kirilovsky A, Berger A, Lagorce C, Paustian C, Ballesteros-Merino C, Dijkstra J, van de Water C, Vliet SVL, Knijn N, Musina AM, Scripcariu DV, Popivanova B, Xu M, Fujita T, Hazama S, Suzuki N, Nagano H, Okuno K, Torigoe T, Sato N, Furuhata T, Takemasa I, Patel P, Vora HH, Shah B, Patel JB, Rajvik KN, Pandya SJ, Shukla SN, Wang Y, Zhang G, Kawakami Y, Marincola FM, Ascierto PA, Fox BA, Pages F, Galon J. Multicenter International Study of the Consensus Immunoscore for the Prediction of Relapse and Survival in Early-Stage Colon Cancer. Cancers (Basel). 2023 Jan 8;15(2):418. doi: 10.3390/cancers15020418. PMID 36672367
- [Background] Pages F, Berger A, Camus M, Sanchez-Cabo F, Costes A, Molidor R, Mlecnik B, Kirilovsky A, Nilsson M, Damotte D, Meatchi T, Bruneval P, Cugnenc PH, Trajanoski Z, Fridman WH, Galon J. Effector memory T cells, early metastasis, and survival in colorectal cancer. N Engl J Med. 2005 Dec 22;353(25):2654-66. doi: 10.1056/NEJMoa051424. PMID 16371631
- [Background] Galon J, Costes A, Sanchez-Cabo F, Kirilovsky A, Mlecnik B, Lagorce-Pages C, Tosolini M, Camus M, Berger A, Wind P, Zinzindohoue F, Bruneval P, Cugnenc PH, Trajanoski Z, Fridman WH, Pages F. Type, density, and location of immune cells within human colorectal tumors predict clinical outcome. Science. 2006 Sep 29;313(5795):1960-4. doi: 10.1126/science.1129139. PMID 17008531
- [Background] Pages F, Kirilovsky A, Mlecnik B, Asslaber M, Tosolini M, Bindea G, Lagorce C, Wind P, Marliot F, Bruneval P, Zatloukal K, Trajanoski Z, Berger A, Fridman WH, Galon J. In situ cytotoxic and memory T cells predict outcome in patients with early-stage colorectal cancer. J Clin Oncol. 2009 Dec 10;27(35):5944-51. doi: 10.1200/JCO.2008.19.6147. Epub 2009 Oct 26. PMID 19858404
- [Background] Mlecnik B, Tosolini M, Kirilovsky A, Berger A, Bindea G, Meatchi T, Bruneval P, Trajanoski Z, Fridman WH, Pages F, Galon J. Histopathologic-based prognostic factors of colorectal cancers are associated with the state of the local immune reaction. J Clin Oncol. 2011 Feb 20;29(6):610-8. doi: 10.1200/JCO.2010.30.5425. Epub 2011 Jan 18. PMID 21245428
- [Background] Mlecnik B, Bifulco C, Bindea G, Marliot F, Lugli A, Lee JJ, Zlobec I, Rau TT, Berger MD, Nagtegaal ID, Vink-Borger E, Hartmann A, Geppert C, Kolwelter J, Merkel S, Grutzmann R, Van den Eynde M, Jouret-Mourin A, Kartheuser A, Leonard D, Remue C, Wang JY, Bavi P, Roehrl MHA, Ohashi PS, Nguyen LT, Han S, MacGregor HL, Hafezi-Bakhtiari S, Wouters BG, Masucci GV, Andersson EK, Zavadova E, Vocka M, Spacek J, Petruzelka L, Konopasek B, Dundr P, Skalova H, Nemejcova K, Botti G, Tatangelo F, Delrio P, Ciliberto G, Maio M, Laghi L, Grizzi F, Fredriksen T, Buttard B, Lafontaine L, Bruni D, Lanzi A, El Sissy C, Haicheur N, Kirilovsky A, Berger A, Lagorce C, Paustian C, Ballesteros-Merino C, Dijkstra J, van de Water C, van Lent-van Vliet S, Knijn N, Musina AM, Scripcariu DV, Popivanova B, Xu M, Fujita T, Hazama S, Suzuki N, Nagano H, Okuno K, Torigoe T, Sato N, Furuhata T, Takemasa I, Itoh K, Patel PS, Vora HH, Shah B, Patel JB, Rajvik KN, Pandya SJ, Shukla SN, Wang Y, Zhang G, Kawakami Y, Marincola FM, Ascierto PA, Fox BA, Pages F, Galon J. Multicenter International Society for Immunotherapy of Cancer Study of the Consensus Immunoscore for the Prediction of Survival and Response to Chemotherapy in Stage III Colon Cancer. J Clin Oncol. 2020 Nov 1;38(31):3638-3651. doi: 10.1200/JCO.19.03205. Epub 2020 Sep 8. PMID 32897827